CLINICAL TRIAL: NCT02890147
Title: Molecular Reclassification to Find Clinically Useful Biomarkers for Systemic Autoimmune Diseases: Case-control
Acronym: PRECISESADST
Status: Completed | Type: Observational
Sponsor: Fundación Pública Andaluza Progreso y Salud (Other)
Collaborators: UCB Biopharma S.P.R.L. (Industry); Atrys Health (Industry); National Research Council, Spain (Other Government); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); Servicio Cántabro de Salud (Other); August Pi Sunyer Biomedical Research Institute (Other); Karolinska Institutet (Other); KU Leuven (Other); Klinikum der Universität Köln (Other); Hannover Medical School (Other); Medical University of Vienna (Other); Quartz Bio S.A. (Other); Andaluz Health Service (Other Government); The Cyprus Foundation for Muscular Dystrophy Research (Other); Universidad de Granada (Other); University of Milan (Other); Université Catholique de Louvain (Other); University Hospital, Brest (Other); University of Geneva, Switzerland (Other); Szeged University (Other); Bayer (Industry); Institut de Recherches Internationales Servier (Other); Sanofi (Industry); Eli Lilly and Company (Industry); Charite University, Berlin, Germany (Other); Centro Hospitalar do Porto (Other); Institut d'Investigació Biomèdica de Bellvitge (Other); Innovative Medicines Initiative (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Other Study IDs: PRECISESADS-T
Record Dates: First submitted 2016-08-22; First posted 2016-09-07 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2018-04

CONDITIONS: Healthy Subjects
Keywords: SADs; Healthy Volunteers; Molecular profiles; Omics Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Connective tissue diseases (CTD) or systemic autoimmune diseases (SADs) as they are known today are a group of chronic inflammatory conditions with autoimmune aetiology with few treatment options and difficult diagnosis.Brest team contribute to perform a new classification of the following systemic autoimmune diseases in a European Union's Seventh Framework Programme. The aim of this research is to constitute a Healthy Volunteers cohort to compare with systemic autoimmune diseases cohort into molecular clusters instead of clinical entities through the determination of molecular profiles using several "Omics" techniques.

DETAILED DESCRIPTION:
The main objective of the PRECISESADS project is to reclassify the individuals affected by SADs into molecular clusters instead of clinical entities through the determination of molecular profiles using several "-omics" techniques.

The specific objectives of this cross sectional study and sub-study are:

1. To identify a systemic taxonomy for patients with SADs by producing the following data in individuals with SADs and controls: genetic, epigenomic, transcriptomic, flow cytometric (from peripheral blood mononuclear and polymorphonuclear cells (PBMCs)), metabolomics and proteomic in plasma and urine, exosome analysis, classical serology (antibodies and autoantibodies), and clinical data.
2. To better characterize individual SADs at the omics level.
3. To perform clustering analyses to determine the groups of individuals who, differentially from other groups, share specific molecular features (precision medicine).
4. To identify gene expression, methylation profiles through deconvolution methods comparing a mixture of cells with subpopulations determined by flow cytometry with separated cells, cytokine profiles and plasma metabolomics using Mass Spectrometry, in a substudy of 288 individuals.

The clustering process will be data-driven with the aim to find the most homogenous and differentiated clusters of diseases that clearly separate individuals on the basis of, serological, genetic, epigenomic, cellular (cell proportions), metabolomic, proteomic (cytokines, autoantibodies) and transcriptome characteristics and differentiate them from controls and other patient clusters.

A total of 2000 patients and 666 controls will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older at the time of consent
* Signed the informed consent form

Exclusion Criteria:

* Individuals on chronic medication.
* Individuals suffering from any inflammatory, autoimmune, allergic or infectious condition and if possible without a history of autoimmune disease, particularly thyroid disease or other diseases that may modify cellular profiles in blood.
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers
Sampling Method: Probability Sample
Enrollment: 649 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Gene expression in total blood | 2 years
  Gene expression will be done using commercial gene expression microarrays in total blood from all samples using the RNA Paxgene tube.
Flow cytometry analysis to determine cell proportions in the total blood mixture in all individuals. | 24 hours
  9 optimized panels of antibodies will be used to determine cell subpopulations in peripheral blood (including very minor cell populations).
Genotyping | 2 years
  Genotyping will be done using a whole genome array.
Metabolite determination | 2 years
  Metabolite determination in plasma and urine using Nuclear Magnetic Resonance
Exosome isolation from plasma and urine | 2 years
  set up of the methodology for isolating exosomes in these bodily fluids for gene expression analysis
Cytokine profile determination | 2 years
  88 different cytokines will be assessed with Luminex
routine autoantibodies in serum | 2 years
  set of serum autoantibodies will be determined in a European validated laboratory. Also, they will perform detection of antibodies against small lipid moieties i.e.antiphosphorylcholine), lupus anticoagulant and complement proteins in plasma.
Gene expression methylation in total blood | 2 years
  Methylation analysis will be done using the methylome 450k array using the DNA obtained from total blood. MicroRNA gene expression arrays using total blood.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Alarcon, Study Director — Fundación Pública Andaluza Progreso y Salud (PHFSpain)
Locations (17):
- Medical University of Vienna, Vienna, Austria
- UZ Leuven - KU Leuven, Department of Rheumatology (KU LEUVEN), Leuven, Belgium
- CHRU de Brest, Brest, France
- Germany (2):
  - Deutsches Rheuma-Forschungszentrum Berlin (DRFZ), Berlin
  - Medizinische Hochschule Hannover, Hanover
- University of Szeged, Szeged, Hungary
- Italy (2):
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico (IRCCS), Milan
  - UNIMI, Istituto Ortopedico Getano Pini, Milan
- Centro Hospitalar do Porto, Porto, Portugal
- Spain (7):
  - Hospital Clinic I Provicia- Institut d'Investigacions Biomèdiques August Pi i Sunyer (IDIBAPS), Barcelona
  - Hospital Universitario Reina Sofía Andaluz de Salud, Córdoba
  - Biobanco del Sistema Sanitario Público de Andalucía (SSPA), Granada
  - Hospital Universitario San Cecilio Servicio Andaluz de Salud, Granada
  - Hospital Virgen de las Nieves Granada, Granada
  - Hospital Regional de Málaga Servicio Andaluz de Salud, Málaga
  - Hospital Universitario Marqués de Valdecilla, Servicio Cántabro de Salud, Santander
- Hospitaux Universitaires de Géneve, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided